CLINICAL TRIAL: NCT04727931
Title: Prevalence of Cognitive Disorders in Newly Diagnosed Epilepsy
Acronym: PRECONISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Maillard Louis, Professor, Central Hospital, Nancy, France
Other Study IDs: n°2020-A00404-35
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Epilepsy; Cognition
Keywords: Newly diagnosed epilepsy; Cognition; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly diagnosed epileptic patients: Newly diagnosed epileptic patients who have never be treated by antiepileptic drugs and who have no psychiatric (mental illness) and/or evolutive neurological history and for minor patients the non-opposition of the parental authority holders.
  Interventions: Behavioral: Neuropsychological assessement and questionnaires
- Normal controls: Matched (on age, gender, socio-educationnal level and manual laterality) healthy controls who have no psychiatric (depression, mental illness) and/or neurological (stroke, traumatic brain injury, etc.) history and for minor patients the non-opposition of the parental authority holders.
  Interventions: Behavioral: Neuropsychological assessement and questionnaires

INTERVENTIONS:
Behavioral: Neuropsychological assessement and questionnaires — Neuropsychological assessement including memory, working memory, executive function, oral naming and speed processing tests. There are questionnaires to assess mood disorders, anxiety and cognitive reserve.

SUMMARY:
A prospective prevalence study recorded that up to 50% of adult patients with newly diagnosed epilepsy had at least one cognitive impairment before initiation of antiepileptic drug (AED). Multiple factors exist and interact in the same patient. Cognitive impairments may affect psychiatric (loss of self-esteem, anxiety, depression) and social status (e.g., vocational aptitude, educational). These factors in turn influence cognitive abilities in a triangular and bidirectional relationship. In addition, the type of epilepsy, development in childhood or cerebral ageing, antiepileptic treatments (AED, surgery) and etiology also have an impact on cognitive performances. The burden of these factors differs from patient to another and must be determined individually. Longitudinal follow-up seems to be crucial because it will allow us to highlight the change in the cognitive profile of newly diagnosed patients over time.

The main objective is to compare the prevalence of cognitive impairment in patients with newly diagnosed epilepsy prior to the initiation of AED with healthy subjects matched on age, sex, manual laterality and socio-educational level. But also to compare the longitudinal evolution of the cognitive profile of patients with healthy controls (0 to 10 years) to determine, among the age of onset seizures, their etiology, the syndrome, the sex, the socio-educational level and the cognitive reserve, which one are related to the severity of cognitive disorders.

ELIGIBILITY:
Inclusion Criteria (patients):

* Individuals who have received full information about the organization of the research and have not refused to participate and to use their data.
* Person aged 16 and over
* For minor patients: the non-opposition of the parental authority holders
* Newly diagnosed epileptic patient who had never taken antiepileptic drugs.

Inclusion Criteria (normal controls):

* Individuals who have received full information about the organization of the research and have not refused to participate and to use their data.
* For minor participants: the non-opposition of the parental authority holders
* Person aged 16 and over.

Exclusion Criteria (patients):

* Person of full age who are subject to a legal protection measure or who are unable to express their consent
* Person with a progressive brain injury
* Person who regularly use psychoactive substances (cannabis, alcohol, etc.)
* Patients who started an antiepileptic treatment before the neuropsychological assessment.

Exclusion Criteria (normal controls):

* Persons of full age who are subject to a legal protection measure or who are unable to express their consent
* Person with a neurological (traumatic brain injury, stroke, etc.) and/or psychiatric (mental illness, depression, etc.) history.
* People who regularly use psychoactive substances (cannabis, alcohol, etc.).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited in the neurology department of the hospital of Nancy. Nomal controls are recruited by display in hospital of Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-02-17 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of impaired cognitive function at the time of diagnosis in patients and healthy subjects. | Baseline (up to 2 weeks after a diagnosis of epilepsy for a duration of 1h30)
  Neuropsychological assessment:
  * BVMT-R
  * RL/RI-16
  * Digit span forward and backward (WASI-IV)
  * Stroop test
  * Verbal fluency
  * TMT
  * Code
  * Oral naming
  Questionnaires:
  * NDDI-E
  * GAD-7
  * Beck inventory
  * STAI
  * CRI-q

SECONDARY OUTCOMES:
Proportion of impaired cognitive functions according to the cognitive domain assessed | Baseline, 6 months, 12 months, 3 years, 6 years and 10 years after the baseline (for a duration of 1h30 at each assessment)
  Participants are assessed 6 times
  Neuropsychological assessment:
  * BVMT-R
  * RL/RI-16
  * Digit span forward and backward (WASI-IV)
  * Stroop test
  * Verbal fluency
  * TMT
  * Code
  * Oral naming
  Questionnaires:
  * NDDI-E
  * GAD-7
  * Beck inventory
  * STAI
  * CRI-q

CONTACTS AND LOCATIONS:
Overall Officials: Louis Maillard, Pr, Principal Investigator — Professor of neurology
Locations (1):
- Department of neurology - Hospital of Nancy, Nancy, France